CLINICAL TRIAL: NCT03042936
Title: Insulin Superheroes Club: Diabetes Prevention Program in Youth (12-month Supplement to the CDC DPP for Adults)
Brief Title: Diabetes Prevention Program in Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-03716-XP
Record Dates: First submitted 2017-01-30; First posted 2017-02-03 (Estimated); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2020-11

CONDITIONS: Pre Diabetes
Keywords: Children; Teens; Adolescents; Type 2 diabetes; Impaired glucose tolerance; Exercise; Nutrition; Education
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Insulin Superheroes Club Curriculum
  Interventions: Behavioral: Insulin Superheroes Club Curriculum

INTERVENTIONS:
Behavioral: Insulin Superheroes Club Curriculum — This curriculum promotes healthier physical activity, nutrition, sleep, and stress coping practices. The intervention lasts 12-months: registration, six evaluation sessions (2-3 hours per evaluation: Weeks 1, 8, and 16, 6-month, 9-month, and 12-month), and 16-weekly, 3-bi weekly, 6-monthly educational and physical activity sessions each lasting 90 minutes.

SUMMARY:
The purpose of this study is to test the effectiveness of an out-of-school diabetes prevention program for youth (ages 7-15) with a family history of pre-diabetes or type 2 diabetes.

DETAILED DESCRIPTION:
The Insulin Superheroes Club (ISC) is based on the Diabetes Prevention Program for adults (Knowler WC et al., 2002), which was developed by the Centers for Disease Control and Prevention (CDC). We have adapted the curriculum for youth to serve a supplement to the adult program. This program lasts 12 months, and the goals are to improve participants' health and reduce their risk of developing pre-diabetes or type 2 diabetes. The ISC program includes 16 weekly (Phase 1), 3 bi-weekly (Phase 2), and 6 monthly (Phase 3) sessions. Sessions include 60 minutes of physical fitness and 30 minutes of education. The education portion includes interactive teaching of a health-related topic (e.g., nutrition, exercise, physiology, mindfulness, and stress reduction) using a hand-on learning activity (e.g., cooking, crafts, games, and role play). All physical fitness activities incorporate moderate intensity exercises (e.g., push-ups, yoga, basketball, tag, and dance).

ELIGIBILITY:
Inclusion criteria

* Between 7-15 years old
* Parent or grandparent with pre/type II Diabetes
* Able to participate in physical activity
* Parent or caregiver participation

Exclusion criteria

* Pregnant females
* Those with significant physical or mental health illness that would hinder study participation
* Medications that would interfere with testing results

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 33 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joan C Han, MD, Principal Investigator — University of Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Derived] Mantilla C, Jones T, Decker KM, Jacobo AM, Sontheimer SY, Mirro MR, Hare ME, Han JC. Diabetes Prevention Program in Youth (Insulin Superheroes Club) Pilot: Improvement in Metabolic Parameters and Physical Fitness After 16 Weeks of Lifestyle Intervention. Diabetes Care. 2017 Jun;40(6):e63-e64. doi: 10.2337/dc16-2678. Epub 2017 Mar 21. No abstract available. PMID 28325785

RESULTS

PARTICIPANT FLOW:
Groups:
- Insulin Superheroes Club Curriculum: A supplement to the Centers for Disease Control and Prevention's adult Diabetes Prevention Program (DPP) designed for youth from culturally diverse, minority backgrounds.
  The ISC is a 12-month, multilevel program that includes 16 weekly (phase 1), 3 biweekly (phase 2), and 6 monthly (phase 3) sessions. Participants attended sessions that included 60 min of physical fitness and 30 min of education. The education portion included interactive teaching of health-related topics (e.g., nutrition, exercise, physiology, mindfulness, and stress reduction) using hands-on learning activities (e.g., cooking, crafts, games, and role-play). All physical fitness activities incorporated moderate-intensity exercises (e.g., push-ups, yoga, basketball, tag, and dance).
Period: Overall Study
Arm/Group | Insulin Superheroes Club Curriculum
Started | 33
Completed | 28
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 33
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.8 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 29
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Hemoglobin A1c
Time Frame: 16 weeks
Measure: Median (Inter-Quartile Range); unit: A1c percentage points
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 33
A1c percentage points | -0.5 [-0.6 to -0.2]

2. Secondary Outcome: Change From Baseline Body Mass Index Z-score
Time Frame: 16 weeks, 6 months, 9 months, 12 months
Population: 0 participants analyzed because data could not be collected.
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 0

3. Secondary Outcome: Change From Baseline Waist Circumference Z-score
Time Frame: 16 weeks, 6 months, 9 months, 12 months
Population: 0 participants analyzed because data could not be collected.
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline Systolic Blood Pressure Z-score
Time Frame: 16 weeks, 6 months, 9 months, 12 months
Population: 0 participants analyzed because data could not be collected.
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 0

5. Secondary Outcome: Change From Baseline Diastolic Blood Pressure Z-score
Time Frame: 16 weeks, 6 months, 9 months, 12 months
Population: 0 participants analyzed because data could not be collected.
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 0

6. Secondary Outcome: Change From Baseline Percent Body Fat
Time Frame: 16 weeks, 6 months, 9 months, 12 months
Population: 0 participants analyzed because data could not be collected.
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 0

7. Secondary Outcome: Change From Baseline Total Cholesterol
Time Frame: 16 weeks, 6 months, 9 months, 12 months
Population: 0 participants analyzed because data could not be collected.
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 0

8. Secondary Outcome: Change From Baseline LDL Cholesterol
Time Frame: 16 weeks, 6 months, 9 months, 12 months
Population: 0 participants analyzed because data could not be collected.
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 0

9. Secondary Outcome: Change From Baseline HDL Cholesterol
Time Frame: 16 weeks, 6 months, 9 months, 12 months
Population: 0 participants analyzed because data could not be collected.
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline Non-HDL Cholesterol
Time Frame: 16 weeks, 6 months, 9 months, 12 months
Population: 0 participants analyzed because data could not be collected.
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 0

11. Secondary Outcome: Change From Baseline Triglycerides
Time Frame: 16 weeks, 6 months, 9 months, 12 months
Population: 0 participants analyzed because data could not be collected.
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 0

12. Secondary Outcome: Change From Baseline Six Minute Walk Test Distance
Time Frame: 16 weeks, 6 months, 9 months, 12 months
Population: 0 participants analyzed because data could not be collected.
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 0

13. Secondary Outcome: Change From Baseline Right Handgrip Strength
Time Frame: 16 weeks, 6 months, 9 months, 12 months
Population: 0 participants analyzed because data could not be collected.
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 0

14. Secondary Outcome: Change From Baseline Left Handgrip Strength
Time Frame: 16 weeks, 6 months, 9 months, 12 months
Population: 0 participants analyzed because data could not be collected.
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 0

15. Secondary Outcome: Change From Baseline Combined Handgrip Strength
Time Frame: 16 weeks, 6 months, 9 months, 12 months
Population: 0 participants analyzed because data could not be collected.
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 0

16. Secondary Outcome: Change From Baseline Sit-and-reach Lower Body Flexibility
Time Frame: 16 weeks, 6 months, 9 months, 12 months
Population: 0 participants analyzed because data could not be collected.
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 0

17. Secondary Outcome: Change From Baseline Shuttle Run Speed
Time Frame: 16 weeks, 6 months, 9 months, 12 months
Population: 0 participants analyzed because data could not be collected.
Arm/Group | Insulin Superheroes Club Curriculum
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Insulin Superheroes Club Curriculum
All-Cause Mortality (participants affected / at risk) | 0/33
Serious Adverse Events (participants affected / at risk) | 0/33
Other Adverse Events (participants affected / at risk) | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-08): https://cdn.clinicaltrials.gov/large-docs/36/NCT03042936/Prot_SAP_000.pdf